CLINICAL TRIAL: NCT04435587
Title: Comparative Efficacy of Ivermectin Versus Combination of Hydroxychloroquine Plus Darunavir/ Ritonavir for Shortening Duration of SARS-CoV2 Detection From Respiratory Secretion Among Asymptomatic or Afebrile COVID-19 Infection
Brief Title: Ivermectin vs Combined Hydroxychloroquine and Antiretroviral Drugs (ART) Among Asymptomatic COVID-19 Infection
Acronym: IDRA-COVID19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Yupin Suputtamongkol, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 323/2563 (IRB3)
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Asymptomatic Infections; SARS-CoV2 Infection
Keywords: ivermectin; hydroxychloroquine/darunavir/ritonavir; SAR-CoV2; asymptomatic infection; zinc sulfate
MeSH Terms: conditions — Asymptomatic Infections; COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: PCR for SAR-CoV2 detection will be performed by technician without knowledge of treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ivermectin (Experimental): Combination of
  1. oral ivermectin 600 mcg/kg/day once daily for 3 days
  2. Zinc sulfate (100mg/tab) 2 tab every 12 hours for 3 days
  Interventions: Drug: Ivermectin Pill
- ART/hydroxychloroquine (Active Comparator): Combination of
  1. Day1 hydroxychloroquine 400mg bid, then 200mg bid on Day 2-5
  2. Darunavir/ritonavir (400/100mg) every 12 hours for 5 days
  3. Zinc sulfate (100/tab) 2 tab every 12 hours for 5 days
  Interventions: Drug: Combined ART/hydroxychloroquine

INTERVENTIONS:
Drug: Ivermectin Pill — 3 days of once daily oral ivermectin 600mcg/kg/d
  Other Names: Vermectin
  Arms: ivermectin
Drug: Combined ART/hydroxychloroquine — 1. Day 1 hydroxychloroquine 400mg bid, Day2-5 hydroxychloroquine 200mg bid
  2. Darunavir/ritonavir (400/100mg) q 12 hours for 5 days
  Other Names: combined darunavir/ritonavir/hydroxychloroquine
  Arms: ART/hydroxychloroquine

SUMMARY:
This is an open label randomised controlled study of oral ivermectin (600 mcg/kg/d* 3 day) versus combined of hydroxychloroquine plus darunavir/ ritonavir for 5 days treatment among asymptomatic carrier of SAR-CoV2 adult Thai population. Both study treatment regimens will have oral zinc sulfate combination treatment ( 200mg. twice daily). Outcomes include safety and duration of detectable of SAR-CoV2 in nasopharyngeal/ throat (NP) swab by polymerase chain reaction amplification (PCR) after treatment. 40-50 patients in each treatment arm is planned, with an interim analysis when approximately 50% of cases is enrolled.

DETAILED DESCRIPTION:
* Study procedure will be carried out after informed consent is obtained.
* Baseline physical exam and laboratory investigations will be performed.
* Eligible patients will be randomized to one of the two treatment arms.
* Symptoms and signs will be monitored daily.
* NP swab will be done at day5-7, and prior to discharge.
* Complete blood counts, blood chemistries, electrocardiography will be performed for adverse event monitoring within 5 days after end of study drugs' administration.
* Patients will be discharged at 2- 4 weeks after hospitalization, according to PCR results.
* There will be 1-2 follow up visit at out patient clinic for NP swab (patients with +ve last NP swab before discharge), and blood tests.
* Additional 5-8 ml. of EDTA blood will be taken at baseline and weekly for antibody detection.
* Interim analysis of both safety and efficacy will be performed when approximately 50% of enrollment is achieved.
* Intention to treat analysis is planned at the completion of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* SAR-CoV2 detected by PCR from NP swab
* Asymptomatic or upper respiratory symptoms such as runny noses
* No history of fever or oral Temp <37.8 degree celsius
* informed consent obtained

Exclusion Criteria:

* Fever or respiratory rate >24/minute or oxygen saturation at room air< 94%
* Any serious co-morbidity such as chronic lung disease, chronic kidney disease, cardiovascular diseases, arrythmia, diabetes mellitus with HbA1C > 8%, chronic liver disease, lymphocyte count <1,000cell/cu.mm.
* History of ivermectin or any of the study drug allergy.
* Concomitant medication with potential drug interaction with any of the study drugs such as alfuzosin, colchicine, ergot derivatives, cisapride, simvastatin and rifampicin
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Adverse event rates | after first dose until day 28 of follow up
  Comparison of adverse event rates between treatment arms
Efficacy for shortening duration of SAR-CoV2 detection by PCR | weekly after treatment until 4th week
  comparison of median duration for detectable SAR-CoV2 by PCR from NP swab in each arm

SECONDARY OUTCOMES:
Antibody detection rates | weekly after treatment until 4th week
  comparison of median duration for total antibody detection in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Yupin Suputtamongkol, MD, Principal Investigator — Department of Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (4):
- Thailand (4):
  - Siriraj Hospital, Bangkok Noi, Bangkok
  - Siriaj Hospital, Bangkok, N/A = Not Applicable
  - Sireethorn Nimitvilai, Amphoe Maueng, Nakhonpathom
  - Golden Jubilee Medical Center, Phutthamonthon District, Nakhonpathom

IPD SHARING:
Plan to Share IPD: No